CLINICAL TRIAL: NCT04150796
Title: Registry Based, Randomized Controlled Trial Comparing eTEP and Laparoscopic Intraperitoneal Onlay Mesh (IPOM) for Ventral Hernia Repair
Brief Title: Comparing eTEP and Laparoscopic Intraperitoneal Onlay Mesh (IPOM) for Ventral Hernias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Clayton Petro, Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-1288
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Ventral Hernia; Umbilical Hernia; Epigastric Hernia
Keywords: Hernia Repair; Minimally-invasive surgery; General surgery
MeSH Terms: conditions — Hernia, Ventral; Hernia, Umbilical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced-view Totally Extraperitoneal (eTEP) Hernia Repair (Experimental): Initial access into the retromuscular space is achieved using an optical trocar. Insufflation of CO2 is performed under direct visualization. Multiple assistant ports will be placed medial to the semilunar line to continue developing the retromuscular space. The medial insertion of the posterior rectus sheath will be incised to enter the preperitoneal plane and facilitate reduction of hernia contents. The contralateral posterior rectus sheath will be incised and the contralateral retrorectus space will be matured. Suture will be used to close any defect in the hernia sac. The defect will be measured, as will be the retrorectus space. The fascial defect will be closed with suture. Non-barrier coated mesh will be placed in the retrorectus space and flat positioning will be confirmed. Ports will be removed under direct visualization, and the abdomen desufflated. Anterior fascia of any larger ports (8mm or greater) will be closed.
  Interventions: Procedure: Ventral Hernia Repair
- Intraperitoneal Onlay Mesh (IPOM) Hernia Repair (Active Comparator): Access is achieved using an optical trocar. Insufflation of CO2 is performed. Two additional trocars are placed on the left side along the anterior axillary line. If necessary, auxiliary ports may be placed on the right side. When present, hernia contents are reduced using graspers. Adhesions between abdominal contents and the abdominal wall are lysed. The hernia defect is identified and measured internally with a sterile plastic ruler with the abdomen insufflated. Defect closure is performed using nonabsorbable suture. Mesh repair is performed using polypropylene mesh with an absorbable hydrogel barrier. Mesh is chosen to achieve a minimum 3 to 5-centimeter overlap from the edges of the closed defect. Inside the abdomen, the mesh is unrolled and positioning against the anterior abdominal wall is confirmed. Mesh edges are fixed circumferentially with permanent fixation. Ports are removed and the abdomen is desufflated. The anterior fascia of the 12mm port is closed.
  Interventions: Procedure: Ventral Hernia Repair

INTERVENTIONS:
Procedure: Ventral Hernia Repair — Participants will undergo robotic ventral hernia repair according to the assigned treatment arm.

SUMMARY:
Ventral hernias can be repaired using a variety of techniques, with smaller defects often being amenable to minimally invasive surgical (MIS) approaches. For many years, the standard of care MIS approach to ventral hernias has been the laparoscopic intraperitoneal onlay mesh (IPOM) approach, in which a large piece of mesh is placed inside of the abdomen and fixed to the inner abdominal wall using a combination of sutures and/or mechanical tacks. For selected patients, the IPOM approach has demonstrated benefits over open repair, including decreased postoperative length of stay and decreased incidence of surgical site infection.

However, concern regarding long-term outcomes of placing mesh inside the abdomen have spurred the search for alternate approaches to MIS ventral hernia repair. This includes the enhanced-view totally extraperitoneal (eTEP) approach, in which the retromuscular plane is accessed and developed so a large piece of mesh may be implanted outside of the abdominal cavity. The theoretical benefits of this approach are that patients may experience reduced pain because mechanical mesh fixation is not required (as compared to traditional IPOM approaches in which mesh is fixed to the inner abdominal wall) and that mesh is kept outside of the abdominal cavity and away from the viscera, allowing use of less expensive, uncoated mesh and theoretically reducing risk for long-term mesh related complications. While popularity of eTEP has grown, literature published regarding this approach has been mostly retrospective, consists of relatively small series of patients, and suffers from selection bias. For the one prospective study of eTEP published by Radu, et al, there was no comparator arm.

The investigators will conduct a registry-based randomized controlled trial comparing MIS approaches for repair of small to medium-sized ventral hernias, specifically eTEP versus IPOM. This will occur through the Americas Hernia Society Quality Collaborative (AHSQC).

Our hypotheses are multiple: 1) Patients with ventral hernias undergoing eTEP will experience a 30% decrease in pain scores by postoperative day 1 compared to patients undergoing IPOM; 2) eTEP will be associated with higher median direct costs per case versus IPOM; 3) eTEP will be associated with equivalent 1-year hernia recurrence rates versus IPOM; 4) eTEP will be associated with significantly increased intraoperative surgeon workload compared to IPOM.

DETAILED DESCRIPTION:
This will be a prospective, registry-based, single-blind, randomized controlled trial with a 1:1 allocation ratio. No important changes to the methods are anticipated. This will be a single-institution study performed at the Cleveland Clinic Foundation in Cleveland, and the AHSQC will serve as our platform for data collection. All enrollments and surgeries in this study will take place at Cleveland Clinic Main Campus.

The study will consist of 2 interventions: IPOM or eTEP. Two expert hernia surgeons with advanced MIS training will enroll patients and perform the operations.

A computer-generated randomization scheme will be built. Randomization will take place on the Research Electronic Data Capture (REDCap®) database program. Patients will be randomized to IPOM or eTEP in the operating room after induction of general anesthesia.

The primary outcome measure is early postoperative pain. Secondary outcome measures are cost, hernia recurrence, and surgeon workload as determined by the NASA Task Load Index (NASA-TLX). The investigators will also collect outcomes pertaining to abdominal wall-specific quality of life (measured by Hernia-Related Quality of Life inventory - HerQLes), and 30-day wound events. No changes to trial outcomes are anticipated, and no interim analyses will be performed. No stopping guidelines are needed, as both eTEP and IPOM represent current standards of care for ventral hernia repair.

Subjects will be blinded to the intervention. A similar number of incisions will be present on the abdomen in similar locations following each intervention, preventing patients from knowing which intervention they received. The investigators are unable to blind the operating surgeon to the intervention arm. The investigators are unable to blind the data collector, the research fellow, to the patients within each intervention arm. However, by utilizing data largely determined from the patients themselves, who will not be informed of the operation that they have received until after study completion, The investigators believe that they are presenting accurate data with limited bias. No subgroup analyses are planned. Patients will not be included for analysis at any time point for which their data is unavailable. Following their 1-year visit, patients will be informed regarding the intervention that they received.

Outcomes to be investigated are based on the study hypotheses and are listed below:

Specific Aim #1: To determine if patients with ventral hernias undergoing eTEP experience a 30% decrease in pain scores by postoperative day 1 compared to patients undergoing IPOM.

The primary outcome is early postoperative pain. Pain will be assessed by Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey and the Numeric Pain Rating Scale (NRS-11). The PROMIS pain intensity 3a survey is a National Institutes of Health developed and validated tool that focuses on patient-reported pain characteristics . The NRS-11 is a frequently utilized pain assessment that consists of an easily administered 0 to 10 Likert scale, in which higher scores reflect greater pain intensity. PROMIS Pain Intensity 3a survey pain scores will be assessed at baseline (at the time of enrollment), at 30 (± 15) and 365 (± 90) days. NRS-11 scores, often used to measure acute pain, will be obtained in the post-anesthesia care unit, and on postoperative days 1 (± 1 days), 7 (± 3 days) and 30 (± 15 days). The NRS-11 scores will be obtained either in person while the patients are hospitalized, or by telephone interview following hospital discharge. Postoperative narcotic requirements, as recorded on standard of care 30-day follow-up forms, will be collected.

Specific Aim #2: To determine if eTEP is associated with higher direct costs compared to IPOM.

A secondary outcome is direct cost at the index surgical admission. Cost data will be obtained from the Cleveland Clinic financial department and will include direct costs. Direct costs for the index operation will include operating room supply and time, intensive care unit, anesthesia, floor care, laboratory tests, radiology and endoscopy, pharmacy, and in-hospital rehabilitation therapies. The operating room supply direct costs for index surgeries will be further categorized into the following groups: mesh and general supply costs. Indirect costs and total charges will be excluded. Capital costs, including the robotic system if used, laparoscopic towers, and non-disposable equipment, will not be included.

Specific Aim #3: To determine if eTEP is associated with equivalent one-year recurrence rates compared to IPOM.

Hernia recurrence will be assessed with the Ventral Hernia Recurrence Inventory survey (VHRI), radiographically, and with clinical exam at 365 (± 90) days. The VHRI, which uses patient-reported outcomes to detect hernia recurrence, is a validated tool that has been shown to detect ventral hernia recurrence with a sensitivity of 85% and a specificity of 81%. If patients do not follow up in person, the VHRI will be applied over the phone by research fellows or coordinators to determine whether hernia recurrence has occurred. If patients follow up in person and have CT scans available, clinical and radiographic assessments of recurrence will be used to determine whether a recurrence has occurred rather than VHRI.

Specific Aim #4: To determine if eTEP is associated with increased intraoperative surgeon workload compared to IPOM.

The investigators plan to measure surgeon workload using the NASA Task Load Index (NASA-TLX) inventory, which is a subjective workload assessment tool for individuals working with human-machine interfaces. This consists of self-reported scales rating an individual's mental demand, physical demand, temporal demand, performance, effort, and frustration. These will be collected from participating surgeons immediately after each operation.

Additional outcomes include abdominal wall-specific quality of life and 30-day wound events. Abdominal wall-specific quality of life will be determined by the HerQLes questionnaire. HerQLes is a 12-question hernia-specific survey that has been previously validated in patients undergoing ventral hernia repair. This will be assessed at baseline, at 30 days (± 15 days) and at 365 days (± 90 days). Wound events are defined as surgical site infection (SSI), surgical site occurrence (SSO) and surgical site occurrences requiring procedural intervention (SSOPI), as defined by the Ventral Hernia Working Group. Wound events will be assessed by a physical exam at 30(± 15) days and 365 (± 90) days. This information is already routinely collected for all patients included in the AHSQC. Additionally, the investigators will plan to obtain yearly follow-up going forward via quality of life surveys and CT scans that are standard of care for our group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Primary ventral or incisional hernia defects
* Midline defect with an expected hernia width equal to or less than 7 centimeters
* Elective hernia repair
* Considered eligible for hernia repair through a minimally-invasive approach
* Able to tolerate general anesthesia
* Able to give consent for participation

Exclusion Criteria:

* Defects greater than 7 centimeters
* Hernia defects considered to require an open approach
* Prior mesh placement in the retrorectus space
* Patients not able to understand and sign a written consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Pain on postoperative day 1 | postoperative day 1
  Pain will be assessed by Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey and the Numeric Pain Rating Scale (NRS-11). The PROMIS pain intensity 3a survey is a National Institutes of Health developed and validated tool that focuses on patient-reported pain characteristics . The NRS-11 is a frequently utilized pain assessment that consists of an easily administered 0 to 10 Likert scale, in which higher scores reflect greater pain intensity.

SECONDARY OUTCOMES:
Pain in post-anesthesia care unit (PACU), on postoperative day 7, at 30-day (15-45 day) follow-up, and at 1-year (9-15 month) follow-up. | immediately postoperatively in post-anesthesia care unit (PACU), on postoperative day 7, at 30-day (15-45 day) follow-up, and at 1-year (9-15 month)
  Pain will be assessed by Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a survey and the Numeric Pain Rating Scale (NRS-11). The PROMIS pain intensity 3a survey is a National Institutes of Health developed and validated tool that focuses on patient-reported pain characteristics . The NRS-11 is a frequently utilized pain assessment that consists of an easily administered 0 to 10 Likert scale, in which higher scores reflect greater pain intensity.
Postoperative narcotic requirements | at 30-day (15-45 day) follow-up
  Patient-reported in morphine equivalent doses (MEDs) on standard of care postoperative survey
Direct costs | index surgical encounter
  Direct costs for the index operation will include operating room supply and time, intensive care unit, anesthesia, floor care, laboratory tests, radiology and endoscopy, pharmacy, and in-hospital rehabilitation therapies. The operating room supply direct costs for index surgeries will be further categorized into the following groups: mesh and general supply costs. Indirect costs and total charges will be excluded.
Hernia recurrence rates | 1 year (9-15 month) follow-up
  Hernia recurrence will be assessed with the Ventral Hernia Recurrence Inventory survey (VHRI), radiographically, and with clinical exam at 365 (± 90) days. The VHRI, which uses patient-reported outcomes to detect hernia recurrence, is a validated tool that has been shown to detect ventral hernia recurrence with a sensitivity of 85% and a specificity of 81%. If patients do not follow up in person, the VHRI will be applied over the phone by research fellows or coordinators to determine whether hernia recurrence has occurred. If patients follow up in person and have CT scans available, clinical and radiographic assessments of recurrence will be used to determine whether a recurrence has occurred rather than VHRI.
Intraoperative Surgeon Workload | index surgery
  We plan to measure surgeon workload using the NASA Task Load Index (NASA-TLX) inventory, which is a subjective workload assessment tool for individuals working with human-machine interfaces. This consists of self-reported scales rating an individual's mental demand, physical demand, temporal demand, performance, effort, and frustration. These will be collected from participating surgeons immediately after each operation.
Abdominal wall-specific quality of life | Baseline, 30-day, 1-year postoperative
  Measured using Hernia-related quality of life survey (HerQLes). This is a scale from 0 to 100 where a higher summary score indicates a better quality of life.
Wound events | at 30(± 15) days and 365 (± 90) days.
  as surgical site infection (SSI), surgical site occurrence (SSO) and surgical site occurrences requiring procedural intervention (SSOPI), as defined by the Ventral Hernia Working Group. Wound events will be assessed by a physical exam at 30(± 15) days and 365 (± 90) days.

CONTACTS AND LOCATIONS:
Overall Officials: Clayton C Petro, MD, Principal Investigator — Assistant Professor of Surgery
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petro CC, Maskal SM, Renton DB, Yunis JP, Meara MP, Diaz K, Wilber M, McKenzie K, Tu C, Phillips SE, Miller BT, Beffa LR, Rosen MJ, Prabhu AS. Robotic Enhanced-View Totally Extraperitoneal vs Intraperitoneal Onlay Mesh Evaluation: 1-Year Exploratory Outcomes of the REVEAL Randomized Clinical Trial. J Am Coll Surg. 2023 Oct 1;237(4):614-620. doi: 10.1097/XCS.0000000000000784. Epub 2023 Jun 13. PMID 37310015